CLINICAL TRIAL: NCT00755417
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Safety and Efficacy of Gabapentin Extended Release (G-ER) Tablets in the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: Study of Gabapentin Extended Release (G-ER) in the Treatment of Vasomotor (Hot Flashes/Hot Flushes) Symptoms in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BREEZE 1; 81-0058
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-02

CONDITIONS: Hot Flashes
Keywords: Hot flashes; Hot flushes; Postmenopausal symptoms; Vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- G-ER 1200 mg (Experimental): Gabapentin extended-release (G-ER) 1200 mg
  Interventions: Drug: Gabapentin Extended-Release (G-ER) 1200 mg
- G-ER 1800 mg (Experimental): Gabapentin extended-release (G-ER) 1800 mg
  Interventions: Drug: Gabapentin Extended-Release (G-ER) 1800 mg
- Sugar Pill (Placebo Comparator): Placebo 1200 mg or 1800 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin Extended-Release (G-ER) 1200 mg — G-ER 1200 mg daily dosage given as two 600-mg tablets.
  Other Names: Gabapentin
  Arms: G-ER 1200 mg
Drug: Gabapentin Extended-Release (G-ER) 1800 mg — G-ER 1800 mg daily dosage given as one 600-mg tablet in the morning and two 600-mg tablets in the evening.
  Other Names: Gabapentin
  Arms: G-ER 1800 mg
Drug: Placebo — Matching placebo dosages of 1200 mg daily (two 600-mg tablets) and 1800 mg daily (one 600-mg tablet in the morning and two 600-mg tablets in the evening).
  Arms: Sugar Pill

SUMMARY:
Depomed's Gabapentin Extended Release (G-ER) is an investigational, extended release formulation of gabapentin that is being studied for the treatment of hot flashes in postmenopausal women.

DETAILED DESCRIPTION:
The primary study objective is to assess the efficacy of G-ER dosed in either of the following regimens:

* G-ER 1200 mg daily (single evening dose)
* G-ER 1800 mg daily (dosed asymmetrically; 600 mg in AM/1200 mg in PM) compared to placebo in reducing the average daily frequency and severity score of moderate to severe hot flashes in postmenopausal women after 4 weeks and 12 weeks of treatment with a stable dose, compared with the baseline week.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women aged 18 to 70 years experiencing ≥7 moderate to severe hot flashes per day (or ≥50 per week) accompanied by sweating during previous 30 days or longer.
2. Had amenorrhea for ≥12 months, amenorrhea for 6 to 12 months with serum follicle-stimulating hormone (FSH) levels >40 mIU/mL, or was ≥6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
3. Willing to discontinue the following: vaginal hormonal products; transdermal or oral estrogen or estrogen/progestin combination; intrauterine progestin; progestin implants; injectable estrogen; topical progesterone cream.
4. Had to have daily average of ≥7 moderate to severe hot flashes and had to complete ≥4 days of diary entries during baseline week to be randomized.
5. If treated with antidepressants, could not have had any changes in drug doses during past month.

Other Inclusions apply.

Exclusion Criteria:

1. Patient treated with a gonadotrophin releasing hormone agonist, anti-estrogens, or aromatase inhibitors within 2 months prior to study entry.
2. Patient treated with estrogen pellets or progestin injectable drugs within 6 months prior to study entry.
3. Patient experience only nighttime hot flashes or worked night shifts on a regular basis.
4. Patient was concurrently treated with gabapentin for other indications. If patient was using gabapentin for treatment of hot flashes, she could be screened after a 7-day washout period provided hot flashes returned.
5. Patient had previously experienced dose-limiting adverse events that prevented titration of gabapentin to an effective dose.
6. Patient had a hypersensitivity to gabapentin.
7. Patient was in an immunocompromised state.
8. Patient had a malignancy other than basal cell carcinoma within 2 years prior to study entry.
9. Patient had gastric reduction surgery, severe chronic diarrhea, chronic constipation, uncontrolled irritable bowel syndrome, uncontrolled inflammatory bowel disease, or unexplained weight loss.
10. Patient had clinically significant abnormal chemistry or hematology results, or calculated glomerular filtration rate <60 mL/min.
11. Patient had history of substance abuse within year prior to study entry.
12. Patient was concurrently taking morphine.
13. Patient had history of chronic hepatitis B or C, hepatitis within 3 months prior to study entry, or history of human immunodeficiency virus.

Other Exclusions apply.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Tempe, Arizona
  - Tucson, Arizona
  - Berkely, California
  - La Mesa, California
  - San Diego, California
  - Santa Rosa, California
  - Denver, Colorado
  - Lakewood, Colorado
  - Waterbury, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Jacksonville, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Sandy Springs, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Madisonville, Kentucky
  - Fall River, Massachusetts
  - Edina, Minnesota
  - St Louis, Missouri
  - Billings, Montana
  - Las Vegas, Nevada
  - Moorestown, New Jersey
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Columbus, Ohio
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Columbia, South Carolina
  - Hilton Head Island, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Bellevue, Washington
  - Renton, Washington
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 541 participants were randomized (enrolled), but only 532 participants received treatment and are included as STARTED.
Period: Overall Study
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Started | 174 (Number of patients that received assigned treatment; ITT and safety populations) | 181 (Number of patients that received assigned treatment; ITT and safety populations) | 177 (Number of patients that received assigned treatment; ITT and safety populations)
Completed | 112 | 126 | 135
Not Completed | 62 | 55 | 42
Not completed — Adverse Event | 28 | 20 | 7
Not completed — Lack of Efficacy | 8 | 4 | 9
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Lost to Follow-up | 3 | 0 | 1
Not completed — Withdrawal by Subject | 12 | 12 | 12
Not completed — Not specified or missing data | 9 | 18 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill | Total
Number analyzed (Participants) | 174 | 181 | 177 | 532
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (5.3) | 52.9 (6.5) | 53.0 (6.6) | 52.9 (6.2)
Age, Customized [Number; unit: Participants]
  <65 years | 170 | 176 | 170 | 516
  >=65 years | 4 | 5 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 181 | 177 | 532
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 121 | 125 | 111 | 357
  Black | 39 | 37 | 50 | 126
  Asian | 1 | 1 | 1 | 3
  Hispanic | 12 | 13 | 12 | 37
  Other | 1 | 5 | 3 | 9
Number of hot flashes in 24-hour period [Mean (Standard Deviation); unit: Hot flashes] — Hot flashes categorized as:
  Mild = sensation of heat without sweating Moderate = sensation of heat with sweating, able to continue activity Severe = sensation of heat with sweating, causing cessation of activity
  Hot flashes
    Moderate hot flashes | 6.1 (4.5) | 6.2 (5.7) | 6.3 (5.6) | 6.2 (5.3)
    Severe hot flashes | 6.4 (4.6) | 7.4 (5.8) | 7.1 (5.9) | 7.0 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Frequency of Hot Flashes After 4 Weeks of Treatment With Daily Doses of G-ER 1200 mg or G-ER 1800 mg Compared to Placebo
Description: Change from baseline in average daily frequency of moderate to severe hot flashes after 4 weeks of treatment with stable daily doses of G-ER 1200 mg or G-ER 1800 mg compared with placebo, using last observation carried forward (LOCF) method of imputation for missing data in intent-to-treat (ITT) population.
Time Frame: From baseline to 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Moderate or severe hot flashes
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 174 | 181 | 177
Moderate or severe hot flashes | -6.8 [-7.37 to -6.13] | -7.3 [-7.89 to -6.71] | -5.8 [-6.41 to -5.18]
Statistical Analysis 1: Comparison: G-ER 1200 mg vs Sugar Pill; Null hypothesis was that there were no treatment differences relative to placebo in mean change from baseline in average daily number of moderate or severe hot flashes at stable dosing Week 4; Test type: Superiority or Other; p = 0.0117, ANCOVA — Based on F test of type III analysis for pairwise comparison at 0.025 level; Included treatment and center factors and baseline value as a covariate, tested at the pairwise 0.025 level; Mean Difference (Final Values) = -0.96, 97.5% CI 2-sided [-1.81 to -0.11], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Based on F test of type III analysis; Included treatment and center factors and baseline value as a covariate, tested at the pairwise 0.025 level; Mean Difference (Final Values) = -1.51, 97.5% CI 2-sided [-2.35 to -0.66], Standard Error of Mean 0.38

2. Primary Outcome: Change From Baseline in Average Daily Frequency of Hot Flashes After 12 Weeks of Treatment With Daily Doses of G-ER 1200 mg or G-ER 1800 mg Compared to Placebo
Description: Change from baseline in average daily frequency of moderate to severe hot flashes after 12 weeks of treatment with stable daily doses of G-ER 1200 mg or G-ER 1800 mg compared with placebo, using last observation carried forward (LOCF) method of imputation for missing data in intent-to-treat (ITT) population.
Time Frame: Form baseline to 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Moderate or severe hot flashes
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 174 | 181 | 177
Moderate or severe hot flashes | -7.4 [-8.10 to -6.73] | -7.4 [-8.04 to -6.74] | -6.9 [-7.53 to -6.18]
Statistical Analysis 1: Comparison: G-ER 1200 mg vs Sugar Pill; Null hypothesis was that there were no treatment differences relative to placebo in mean change from baseline in average daily number of moderate or severe hot flashes at stable dosing Week 12; Test type: Superiority or Other; p = 0.1830, ANCOVA — Based on F test of type III analysis; Included treatment and center factors and baseline value as a covariate, tested at the pairwise 0.025 level; Mean Difference (Final Values) = -0.56, 97.5% CI 2-sided [-1.49 to 0.38], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1975, ANCOVA — Based on F test of type III analysis; Included treatment and center factors and baseline value as a covariate, tested at the pairwise 0.025 level; Mean Difference (Final Values) = -0.53, 97.5% CI 2-sided [-1.46 to 0.40], Standard Error of Mean 0.41

3. Primary Outcome: Change From Baseline in Average Daily Severity Score of Hot Flashes After 4 Weeks of Treatment With Daily Doses of G-ER 1200 mg or G-ER 1800 mg Compared to Placebo
Description: Change from baseline in average daily severity score of moderate to severe hot flashes after 4 weeks of treatment with stable daily doses of G-ER 1200 mg or G-ER 1800 mg compared with placebo, using last observation carried forward (LOCF) method of imputation for missing data in intent-to-treat (ITT) population. Severity score is on a 3-point scale where 1=Mild, 2=Moderate, and 3=Severe.
Time Frame: From baseline to 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a numerical scale
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 174 | 181 | 177
Score on a numerical scale | -0.5 [-0.68 to -0.41] | -0.6 [-0.74 to -0.48] | -0.3 [-0.42 to -0.15]
Statistical Analysis 1: Comparison: G-ER 1200 mg vs Sugar Pill; Null hypothesis was that there were no treatment differences relative to placebo in mean change from baseline in average daily severity score of moderate or severe hot flashes at stable dosing Week 4; Test type: Superiority or Other; p = 0.0016, ANCOVA — Based on F test of type III analysis; Included treatment and center factors and baseline value as a covariate, tested at the pairwise 0.025 level; Mean Difference (Final Values) = -0.26, 97.5% CI 2-sided [-0.44 to -0.08], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Based on the F test of type III analysis; Included treatment and center factors and baseline value as a covariate, tested at the pairwise 0.025 level; Mean Difference (Final Values) = -0.32, 97.5% CI 2-sided [-0.51 to -0.14], Standard Error of Mean 0.08

4. Primary Outcome: Change From Baseline in Average Daily Severity Score of Hot Flashes After 12 Weeks of Treatment With Daily Doses of G-ER 1200 mg or G-ER 1800 mg Compared to Placebo
Description: Change from baseline in average daily severity score of moderate to severe hot flashes after 12 weeks of treatment with stable daily doses of G-ER 1200 mg or G-ER 1800 mg compared with placebo, using last observation carried forward (LOCF) method of imputation for missing data in intent-to-treat (ITT) population. Severity score is on a 3-point scale were 1=Mild, 2=Moderate, and 3=Severe.
Time Frame: From baseline to 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a numerical scale
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Number analyzed (Participants) | 174 | 181 | 177
Score on a numerical scale | -0.7 [-0.91 to -0.58] | -0.7 [-0.90 to -0.59] | -0.5 [-0.71 to -0.38]
Statistical Analysis 1: Comparison: G-ER 1200 mg vs Sugar Pill; Null hypothesis was that there were no treatment differences relative to placebo in mean change from baseline in average daily severity score of moderate or severe hot flashes at stable dosing Week 12; Test type: Superiority or Other; p = 0.0433, ANCOVA — Based on the F test of type III analysis; Included treatment and center factors and baseline value as a covariate, tested at the pairwise 0.025 level; Mean Difference (Final Values) = -0.20, 97.5% CI 2-sided [-0.43 to 0.02], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: G-ER 1800 mg vs Sugar Pill; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0468, ANCOVA — Based on the F test of type III analysis; Included treatment and center factors and baseline value as a covariate, tested at the pairwise 0.025 level; Mean Difference (Final Values) = -0.20, 97.5% CI 2-sided [-0.42 to 0.03], Standard Error of Mean 0.10

ADVERSE EVENTS:
Time Frame: Total of 26 weeks: from randomization through 1 week after study completion (week 25).
Description: Adverse events that occurred when patient signed informed consent form through completion of 1-week follow-up telephone contact after end-of-treatment visit at week 25 (stable dosing week 24).
Arm/Group | G-ER 1200 mg | G-ER 1800 mg | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 2/174 | 6/181 | 4/177
Other Adverse Events (participants affected / at risk) | 148/174 | 167/181 | 65/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-ER 1200 mg (N=174) | G-ER 1800 mg (N=181) | Sugar Pill (N=177)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease exacerbation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-ER 1200 mg (N=174) | G-ER 1800 mg (N=181) | Sugar Pill (N=177)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 9 (9)
Dizziness (Nervous system disorders) | 41 (41) | 35 (35) | 5 (5)
Fatigue (General disorders) | 9 (9) | 9 (9) | 3 (3)
Flatulence (Gastrointestinal disorders) | 11 (11) | 7 (7) | 2 (2)
Headache (Nervous system disorders) | 15 (15) | 17 (17) | 10 (10)
Nasopharyngitis (Infections and infestations) | 14 (14) | 11 (11) | 7 (7)
Nausea (Gastrointestinal disorders) | 12 (12) | 16 (16) | 7 (7)
Somnolence (Nervous system disorders) | 23 (23) | 35 (35) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 10 (10) | 10 (10)
Vomiting (Gastrointestinal disorders) | 3 (3) | 13 (13) | 4 (4)
Weight increased (Investigations) | 5 (5) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agree that the sponsor shall have the right to the first publication of the results of the study which is intended to be joint, multi-center publication. Following the first publication, the PI may publish data or results from the study, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the data of the proposed publication.Sponsor may remove any information that is considered confidential and or proprietary other than study data.